CLINICAL TRIAL: NCT01894243
Title: An Open-label, Non-randomised, Multicentre, Comparative, Phase I Study to Determine the Pharmacokinetics, Safety and Tolerability of Olaparib Following a Single Oral 300 mg Dose to Patients With Advanced Solid Tumours and Normal Hepatic Function or Mild or Moderate Hepatic Impairment
Brief Title: Study to Assess the Blood Levels and Safety of Olaparib in Patients With Advanced Solid Tumours and Normal Liver Function or Mild or Moderate Liver Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D0816C00005; 2013-002246-37 (EudraCT Number)
Record Dates: First submitted 2013-07-04; First posted 2013-07-10 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-07

CONDITIONS: Solid Tumours
Keywords: oncology,; cancer,; neoplasm,; anticancer drug,; pharmacokinetics,; area under curve,; olaparib,; solid tumour,; mild hepatic impairment,; moderate hepatic impairment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal hepatic function (Other): Patients with:
  (i) negative result for serum hepatitis B surface antigen and hepatitis C antibody (ii) total bilirubin ≤1.5 x institutional upper limit of normal (ULN), albumin and prothrombin time within normal limits and must not have ascites (unless related to disease under study) or encephalopathy (iii) aspartate aminotransferase or serum glutamic oxaloacetic transaminase (AST), alanine aminotransferase or serum glutamic pyruvic transaminase (ALT) ≤2.5 x institutional ULN unless liver metastases are present in which case it must be ≤5 x ULN
  Interventions: Drug: Olaparib tablet dosing
- Mild hepatic impairment (Other): As defined by the Child-Pugh Classification System.
  Interventions: Drug: Olaparib tablet dosing
- Moderate hepatic impairment (Other): As defined by the Child-Pugh Classification System.
  Interventions: Drug: Olaparib tablet dosing

INTERVENTIONS:
Drug: Olaparib tablet dosing — Part A - single 300mg oral dose olaparib (administered as 2x150mg tablets) Part B - 300mg oral dose olaparib (administered as 2x150mg tablets) bd

SUMMARY:
This is a 2-part study in patients with advanced solid tumours. Part A will investigate the PK of olaparib in patients with mild or moderate hepatic impairment compared to patients with normal hepatic function; Part B will allow patients with mild or moderate hepatic impairment or normal hepatic function continued access to olaparib after the PK phase and will provide additional safety data.

ELIGIBILITY:
Inclusion criteria:-

For inclusion in the study as a patient with hepatic impairment, the following criterion must be met:

1. Patients must have stable mild hepatic impairment (as defined by Child-Pugh classification), for at least 1 month prior to the start of the study or stable moderate hepatic impairment ( as defined by Child Pugh classification) for at least 2 weeks prior to the start of the study. Patients with hepatic metastases and/or HCC are eligible for the study, providing the hepatic metastases or HCC are not the sole reason for any changes in liver function satisfying the criteria for mild or moderate hepatic impairment as defined by the Child Pugh criteria. Patients must have globally impaired hepatic function to participate in the study. For inclusion in the study as a patient with normal hepatic function, the following criteria must be met:
2. Negative result for serum hepatitis B surface antigen and hepatitis C antibody.
3. Total bilirubin less than or equal to1.5 x institutional upper limit of normal (ULN), albumin and prothrombin time within normal limits and must not have ascites (unless related to disease under study) or encephalopathy.
4. Aspartate aminotransferase or serum glutamic oxaloacetic transaminase (AST), alanine aminotransferase or serum glutamic pyruvic transaminase (ALT) less than or equal to 2.5 x institutional ULN unless liver metastases are present in which case it must be less than or equal to 5 x ULN. All patients must fulfil the following criteria:
5. Provision of written informed consent prior to any study specific procedures.
6. Patients must be greater than or equal to18 years of age.
7. Histologically or, where appropriate, cytologically confirmed malignant solid tumour refractory or resistant to standard therapy or for which no suitable effective standard therapy exists. In case of HCC, histological or cytological confirmation is not required in the following situations, as per international guidelines of the scientific societies European Society for Medical Oncology (ESMO) and

   American Association for the Study of Liver Diseases (AASLD):
   * Nodules >2 cm with a typical feature of HCC on a dynamic imaging technique, or any nodule associated with α-fetoprotein (AFP) concentration >400 ng/ml or rising AFP on sequential determinations, do not require biopsy but should be considered as proven HCC (Jelic et al 2010).
   * Nodules >1 cm found on ultrasound screening of a cirrhotic liver should be investigated further with either 4-phase multi-detector CT scan or dynamic contrast enhanced MRI. If the appearances are typical of HCC (ie, hyper-vascular in the arterial phase with washout in the portal venous or delayed phase), the lesion should be treated as HCC. If the findings are not characteristic or the vascular profile is not typical, a second contrastenhanced study with the other imaging modality should be performed, or the lesion should be biopsied (level II) (Bruix et al 2011).
8. Normal organ and bone marrow function measured within 28 days prior to administration of IP as defined below: Haemoglobin greater than or equal to 9.0 g/dL, with no blood transfusions in the previous 28 days.

   Absolute neutrophil count (ANC) greater than or equal to1.5 x 109/L. White blood cells (WBC) greater than 3 x 109/L. Platelet count greater than or equal to 75 x 109/L. Serum creatinine less than or equal to1.5 x institutional ULN.
9. Calculated serum creatinine clearance greater than 50 mL/min (using Cockcroft-Gault formula or by 24-hour urine collection).
10. Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
11. Patients must have a life expectancy greater than or equal to 8 weeks.
12. Evidence of non childbearing status for women of childbearing potential, or postmenopausal status: negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on Day 1 of the first treatment period in Part A. Postmenopausal is defined as:

    Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments.

    Luteinising hormone and follicle-stimulating hormone levels in the postmenopausal range for women under 50 years of age.

    Radiation-induced oophorectomy with last menses greater than 1 year ago. Chemotherapy-induced menopause with greater than 1 year interval since last menses.

    Surgical sterilisation (bilateral oophorectomy or hysterectomy).
13. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
14. Patients must be on a stable concomitant medication regimen (with the exception of electrolyte supplements), defined as no changes in medication or in dose within 2 weeks prior to start of olaparib dosing, except for bisphosphonates, denosumab and corticosteroids, which should be stable for at least 4 weeks prior to start of olaparib dosing.

Exclusion criteria:-

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff, its agents and/or staff at the study site).
2. Previous enrolment in the present study.
3. Treatment with any investigational product (IP) during the last 14 days (or a longer period depending on the defined characteristics of the agent used).
4. Treatment in the previous 3 months before dosing in this study with any drug known to have a well defined potential for hepatoxicity (eg, halothane).
5. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 2 weeks prior to study treatment. The patient can receive a stable dose of bisphosphonates or denosumab for bone metastases before and during the study as long as these were started at least 4 weeks prior to treatment.
6. Patients who have received or are receiving inhibitors or inducers of CYP3A4 within the washout period.
7. Toxicities (greater than or equal to CTCAE Grade 2) caused by previous cancer therapy, excluding alopecia.
8. Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. Patients with asymptomatic brain metastases or with symptomatic but stable brain metastases can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment.
9. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of major surgery.
10. Patients considered a poor medical risk due to a serious uncontrolled medical disorder, non malignant systemic disease, uncontrolled seizures, or active uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive bilateral interstitial lung disease on high resolution computer tomography (HRCT) scan, or any psychiatric disorder that prohibits obtaining informed consent.
11. Patients with a history of heart failure or left ventricular dysfunction.

2. Patients who have gastric, gastro-oesophageal or oesophageal cancer. 13. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders or significant gastrointestinal resection likely to interfere with the absorption of olaparib.

14. Breastfeeding women. 15. Immunocompromised patients eg, patients who are known to be serologically positive for human immunodeficiency virus (HIV).

16. Patients with a known hypersensitivity to olaparib or any of the excipients of the product. 17. Resting ECG with measurable QTc greater than 470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.

18. Clinical judgment by the investigator that the patient should not participate in the study. In addition to exclusion criteria 1 to 18, patients with normal hepatic function should not enter the study if the following exclusion criterion is fulfilled: 19. History or presence of hepatic disease known to interfere with the absorption, distribution, metabolism or excretion of olaparib. In addition to exclusion criteria 1 to 18, patients with mild or moderate hepatic impairment should not enter the study if the following exclusion criteria are fulfilled: 20. Patients with hepatic encephalopathy (as described in the Child Pugh Classification system).

21. Fluctuating or rapidly deteriorating hepatic function as indicated by widely varying or worsening of clinical and/or laboratory signs of hepatic impairment within the screening period (eg, advanced ascites, fever, active gastrointestinal bleeding).

22. Change in dose regimen of medically required medication within the last 2 weeks before screening and/or the use of disallowed co-medication in the 3 weeks prior to admission to the clinic.

23. Presence of acute liver disease caused by drug toxicity or by an infection. 24. Severe portal hypertension or surgical porto-systemic shunts. 25. Biliary obstruction or other causes of hepatic impairment not related to parenchymal disorder and/or disease of the liver.

26. Oesophageal variceal bleeding within the past 2 months. 27. Anticoagulant therapy with warfarin or related coumarins.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-03-13 (Actual); Primary Completion 2016-11-29 (Actual); Study Completion 2017-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anitra Fielding, Study Director — AstraZeneca Senior Research Physician; Christian Rolfo, Principal Investigator — UZ Antwerpen
Locations (11):
- Research Site, Brno, Czechia
- France (5):
  - Research Site, Bordeaux
  - Research Site, Dijon
  - Research Site, Grenoble
  - Research Site, Lyon
  - Research Site, Paris
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Maastricht
- Research Site, Seoul, South Korea
- United Kingdom (2):
  - Research Site, London
  - Research Site, Sutton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled on 13 March 2014 and the last patient was enrolled on 23 January 2015. Patients were enrolled at 8 centers in 3 countries. Of the 31 patients enrolled, 24 were assigned to treatment.
Pre-assignment Details: Approximately 30 patients were planned to be enrolled with at least 24 evaluable patients required to complete Part A (8 patients with normal hepatic function, 8 with mild hepatic impairment and 8 with moderate hepatic impairment). An evaluable patient is defined as a patient having full PK sampling to 96 hours post-dose of olaparib
Groups:
- Normal Hepatic Function: Olaparib 300 mg (2x150 mg tablets) single dose administered to patients with normal hepatic function
- Mild Hepatic Impairment: Olaparib 300 mg (2x150 mg tablets) single dose administered to patients with mild hepatic function
- Moderate Hepatic Impairment: Olaparib 300 mg (2x150 mg tablets) single dose administered to patients with moderate hepatic function
Period: Overall Study
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Started (Received treatment in Part A) | 13 | 10 | 8
Completed Treatment in Part A | 13 | 10 | 8
Ongoing Into Part B | 13 | 10 | 8
Completed (Completed treatment in Part B) | 0 | 0 | 0
Not Completed | 13 | 10 | 8
Not completed — Adverse Event | 0 | 1 | 2
Not completed — Death | 0 | 0 | 3
Not completed — Lack of Efficacy | 3 | 3 | 1
Not completed — Condition under investigation worsened | 8 | 6 | 2
Not completed — Subject decision | 1 | 0 | 0
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Total
Number analyzed (Participants) | 13 | 10 | 8 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (8.35) | 57.4 (10.70) | 67.9 (9.22) | 56.8 (9.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 2 | 14
  Male | 5 | 6 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: Summary of Geometric Least Squares (GLS) Mean for normal, mild and moderate hepatic impairment
Time Frame: Blood samples are collected at pre-dose, 0.25 , 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours post olaparib dose in Part A.
Population: PK Analysis Set (Part A) One patient excluded from mild impairment arm due to surgery that may affect olaparib absorption.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: μg/mL
Groups:
- Moderate Hepatic Function: Olaparib 300 mg (2x150 mg tablets) single dose administered to patients with moderate hepatic function
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Function
Number analyzed (Participants) | 13 | 9 | 8
μg/mL | 7.32 [5.95 to 9.00] | 8.25 [6.43 to 10.58] | 6.40 [4.92 to 8.34]

2. Primary Outcome: Ratio of Maximum Plasma Concentration (Cmax) - Mild vs Normal and Moderate vs Normal
Description: Summary of ratio of Geometric Least Squares (GLS) Means
Time Frame: as for outcome 1
Population: PK Analysis Set (Part A) One patient excluded from mild impairment group due to surgery that may affect olaparib absorption.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Groups:
- GLSMean Ratio of Mild to Normal: Olaparib 300 mg (2x150 mg tablets) single dose administered to patients with mild/normal hepatic function
- GLSMean Ratio of Moderate to Normal: Olaparib 300 mg (2x150 mg tablets) single dose administered to patients with moderate/normal hepatic function
Arm/Group | GLSMean Ratio of Mild to Normal | GLSMean Ratio of Moderate to Normal
Number analyzed (Participants) | 22 | 21
ratio | 1.13 [0.82 to 1.56] | 0.87 [0.63 to 1.22]

3. Primary Outcome: Area Under the Plasma Concentration Time Curve From Zero to Infinity (AUC)
Description: Summary of Geometric Least Squares (GLS) Mean
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: μg*h/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 13 | 9 | 8
μg*h/mL | 52.33 [38.88 to 70.43] | 60.25 [42.17 to 86.10] | 56.29 [38.55 to 82.20]

4. Primary Outcome: Ratio of Area Under the Plasma Concentration Time Curve From Zero to Infinity (AUC) - Mild vs Normal and Moderate vs Normal
Description: Summary of Ratio of Geometric Least Squares (GLS) Means
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | GLSMean Ratio of Mild to Normal | GLSMean Ratio of Moderate to Normal
Number analyzed (Participants) | 22 | 21
ratio | 1.15 [0.72 to 1.83] | 1.08 [0.66 to 1.74]

5. Primary Outcome: Area Under the Plasma Concentration Time Curve From Zero to the Last Measureable Time Point(AUC 0-t)
Description: Summary of Geometric Least Squares (GLS) Mean for ratio of mild hepatic impairment compared to normal
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: μg*h/mL
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Function
Number analyzed (Participants) | 13 | 9 | 8
μg*h/mL | 51.82 [38.69 to 69.40] | 59.64 [41.99 to 84.73] | 55.97 [38.57 to 81.22]

6. Primary Outcome: Ratio of Area Under the Plasma Concentration Time Curve From Zero to the Last Measureable Time Point(AUC 0-t)
Description: Summary of Ratio of Geometric Least Squares (GLS) Means
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | GLSMean Ratio of Mild to Normal | GLSMean Ratio of Moderate to Normal
Number analyzed (Participants) | 22 | 21
ratio | 1.15 [0.73 to 1.82] | 1.08 [0.67 to 1.73]

7. Primary Outcome: Apparent Clearance Following Oral Administration (CL/F)
Description: Summary of Geometric Least Squares (GLS) Means
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: L/hr
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 13 | 9 | 8
L/hr | 5.73 [4.26 to 7.72] | 4.98 [3.48 to 7.11] | 5.33 [3.65 to 7.78]

8. Primary Outcome: Ratio of Apparent Clearance Following Oral Administration (CL/F)
Description: Summary of Ratio of Geometric Least Squares (GLS) Means
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Groups:
- GLSMean Ration of Mild to Normal: Olaparib 300 mg (2x150 mg tablets) single dose administered to patients with mild/normal hepatic function
Arm/Group | GLSMean Ration of Mild to Normal | GLSMean Ratio of Moderate to Normal
Number analyzed (Participants) | 22 | 21
ratio | 0.87 [0.55 to 1.38] | 0.93 [0.57 to 1.50]

9. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax)
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: h
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 13 | 9 | 8
h | 1.53 [0.93 to 6.00] | 2.05 [1.50 to 6.08] | 1.54 [0.50 to 6.00]

10. Primary Outcome: Terminal Half-life (t½)
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 13 | 9 | 8
h | 17.41 (61.7) | 16.58 (49.6) | 13.70 (37.5)

11. Primary Outcome: Apparent Volume of Distribution (Vz/F)
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment
Number analyzed (Participants) | 13 | 9 | 8
L | 144.0 (62.5) | 119.1 (58.7) | 105.4 (84.0)

ADVERSE EVENTS:
Time Frame: Onset date between the date of first dose in Part A and the day before first dose in Part B, or 30 days following the date of last dose of study medication if the subject has discontinued in Part A. For Part B, onset date on or after the first dose in Part B, and up to (and including) 30 days after the last dose date in the study.
Groups:
- Normal (Part A): Normal hepatic function (Part A)
- Mild (Part A): Mild hepatic impairment (Part A)
- Moderate (Part A): Moderate hepatic impairment (Part A)
- Normal (Part B): Normal hepatic function
- Mild (Part B): Mild hepatic impairment (Part B)
- Moderate (Part B): Moderate hepatic impairment (Part B)
Arm/Group | Normal (Part A) | Mild (Part A) | Moderate (Part A) | Normal (Part B) | Mild (Part B) | Moderate (Part B)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/10 | 0/8 | 1/13 | 1/10 | 4/8
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/10 | 1/8 | 3/13 | 3/10 | 4/8
Other Adverse Events (participants affected / at risk) | 10/13 | 3/10 | 5/8 | 13/13 | 10/10 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal (Part A) (N=13) | Mild (Part A) (N=10) | Moderate (Part A) (N=8) | Normal (Part B) (N=13) | Mild (Part B) (N=10) | Moderate (Part B) (N=8)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Normal (Part A) (N=13) | Mild (Part A) (N=10) | Moderate (Part A) (N=8) | Normal (Part B) (N=13) | Mild (Part B) (N=10) | Moderate (Part B) (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 7 (7) | 5 (5) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0/1 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days